CLINICAL TRIAL: NCT03235739
Title: Ancillary Effects of Oral Naloxegol (Movantik)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Alparslan Turan, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-765
Record Dates: First submitted 2017-07-18; First posted 2017-08-01 (Actual); Results first posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — naloxegol

STUDY DESIGN:
Intervention Model Description: Effect of Naloxegol on reversing opioid-related side effects in patients recovering from elective primary hip surgery under spinal anesthesia who will be randomly assigned to oral Naloxegol or placebo for two postoperative days or until the date of discharge, whichever occurs earlier. The design will be a randomized, double-blind, placebo-controlled trial of oral Naloxegol in adults having elective primary hip or knee surgery under spinal anesthesia. The study will be performed at the Cleveland Clinic hospitals.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Naloxegol 25 mg given once in the morning every day until Post-operative Day 3 or day of discharge whichever occurs first
  Interventions: Drug: Naloxegol 25 MG
- Placebo Arm (Placebo Comparator): Matching placebo given once in the morning every day until Post-operative Day 3 or day of discharge whichever occurs first
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naloxegol 25 MG — Oral Naloxegol 25 MG
  Other Names: Movantik
  Arms: Treatment Arm
Drug: Placebo — matching oral placebo
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to find out whether oral Naloxegol can reduce the side effects of opioid painkillers following surgery. This study aims to explore whether Naloxegol can similarly reduce opioid-induced side effects in post-surgical patients. About 130 surgery patients will participate in this study which is being conducted at Cleveland Clinic Main Campus.

DETAILED DESCRIPTION:
Opioids are the gold standard for postoperative pain management, but they have been shown to produce uncomfortable side effects such as urinary retention (an inability to completely empty the bladder), constipation and nausea/vomiting. Clinical evidence demonstrates that Naloxegol can safely and effectively block these undesirable side effects while maintaining the painkilling effects of opioids in outpatients suffering from opioid-induced constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female or male aged at least 18 years
3. American Society of Anesthesiologists physical status 1-4;
4. Scheduled for elective primary hip or knee surgery under spinal anesthesia;
5. Expected to receive intravenous patient-controlled analgesia (IV PCA)
6. Expected to have significant postoperative pain
7. Negative pregnancy test

Exclusion Criteria:

1. Severe hepatic impairment, with/or twice the upper normal levels of liver enzymes
2. Severe renal impairment, or creatinine level > 2.0
3. History of bladder cancer
4. Patients receiving perioperative regional anesthesia blocks
5. Presence of a sacral nerve stimulator
6. Medications (anticholinergic agents such as antihistamines, phenothiazines, antidepressants, antipsychotics), conditions or comorbidity causing urinary retention
7. Patient with requirement of urinary catheter insertion before or immediately post-surgery due to immobility
8. Urinary Tract Infections and other urogenital comorbidity (incontinence, cysto-ureteric reflux, known bladder retention) or conditions which can cause urinary retention
9. Severe peptic ulcer disease, diverticular disease, infiltrative gastrointestinal tract malignancies, or peritoneal metastases
10. Patients with known or suspected disruption of blood brain barrier, which may include but not limited to: Alzheimer's disease, stroke, poliomyelitis, cerebral palsy, multiple sclerosis, spinal lesions, and Parkinson's disease
11. Gastrointestinal obstruction/Gastrointestinal perforation
12. Strong CYP3A4 inhibitors (some antibiotics, antifungals, protease inhibitors, and antidepressants), Strong CYP3A4 inducers, Other opioid antagonists
13. Hypersensitivity to MOVANTIK (naloxegol) or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet A Turan, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data to be provided in aggregate without patient identifiers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: of 508 patients screened, 136 patients meet all inclusion and exclusion criteria and gave consent to the study. 136 patients were randomized.
Groups:
- Treatment-Naloxegol: Naloxegol 25 mg given once in the morning every day until Post-operative Day 3 or day of discharge whichever occurs first
  Naloxegol 25 MG: Oral Naloxegol 25 MG
Period: Overall Study
Arm/Group | Treatment-Naloxegol | Placebo Arm
Started | 69 | 67
Completed | 67 | 64
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment-Naloxegol | Placebo Arm | Total
Number analyzed (Participants) | 67 | 64 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (13) | 62 (11) | 63 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 35 | 32 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 59 | 57 | 116
  African American | 6 | 5 | 11
  Other | 1 | 0 | 1
  Unknown | 1 | 2 | 3
ASA status [Count of Participants; unit: Participants] — ASA Physical Status Classification System, where lower number means better condition. I means a normal healthy patient and VI means a declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    1 | 1 | 1 | 2
    2 | 8 | 15 | 23
    3 | 52 | 46 | 98
    4 | 6 | 2 | 8
Apfel PONV score [Median (Inter-Quartile Range); unit: units on a scale] — Apfel Score for Postoperative Nausea and Vomiting. The EMR- based risk scoring tool was integrated into all preanesthetic assessments and allowed for the assignment of low, moderate, or high risk of PONV. Low risk was defined as an Apfel score of 0 to1, medium risk was defined as an Apfel score of 2, and high risk was defined as an Apfel score of 3 or greater. The minimum of the score is 0 and maximum score is 4.
  units on a scale | 2 [2 to 3] | 2 [2 to 3] | 2 [2 to 3]
Chronic opioid use [Count of Participants; unit: Participants] — Chronic opioid use will be defined as opioid use for more than 30 consecutive days, at a daily dose of 15 mg or more of morphine or equivalent, within the 3 months before surgery.
  Participants | 36 | 32 | 68
Surgery type [Count of Participants; unit: Participants]
  Hip | 67 | 64 | 131
  Knee | 0 | 0 | 0
Surgery duration [Median (Inter-Quartile Range); unit: hours] | 3.6 [2.9 to 4.7] | 3.5 [2.9 to 4.5] | 3.6 [2.9 to 4.5]
Medical history [Count of Participants; unit: Participants]
  Kidney disease | 4 | 1 | 5
  chronic pulmonary disease | 9 | 9 | 18
  obstructive sleep apnea | 9 | 6 | 15
  diabetes mellitus | 7 | 7 | 14
  myocardial infarction | 6 | 4 | 10
  Ischemic Heart Disease | 14 | 10 | 24
  neurological disease | 7 | 12 | 19
  chronic pain | 1 | 5 | 6
  current smoker | 9 | 7 | 16
  drug user | 2 | 5 | 7
  alcohol abuse | 10 | 7 | 17
  cancer | 10 | 6 | 16
Anesthesia type [Count of Participants; unit: Participants] — Population: one patient was missing on anesthesia type information
  Participants
    number analyzed (Participants) | 67 | 63 | 130
    General anesthesia | 46 | 45 | 91
    Spinal anesthesia | 21 | 18 | 39
Intraoperative colloids, ml [Median (Inter-Quartile Range); unit: ml] — Population: one patient was missing on colloids information
  ml
    number analyzed (Participants) | 67 | 63 | 130
    (all) | 0 [0 to 500] | 0 [0 to 250] | 0 [0 to 300]
Intraoperative crystalloids [Median (Inter-Quartile Range); unit: ml] — Population: one patient was missing on crystalloids
  ml
    number analyzed (Participants) | 67 | 63 | 130
    (all) | 2000 [1400 to 2700] | 1800 [1400 to 2700] | 1900 [1400 to 2700]
Intraoperative RBC [Median (Inter-Quartile Range); unit: cc] — Population: one patient was missing
  cc
    number analyzed (Participants) | 67 | 63 | 130
    (all) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Intraoperative platelets [Median (Inter-Quartile Range); unit: cc] — Population: one patient was missing
  cc
    number analyzed (Participants) | 67 | 63 | 130
    (all) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
intraoperative Urine [Median (Inter-Quartile Range); unit: cc] — Population: one patient was missing
  cc
    number analyzed (Participants) | 67 | 63 | 130
    (all) | 0 [0 to 420] | 0 [0 to 460] | 0 [0 to 420]
Intraoperative opioid use [Median (Inter-Quartile Range); unit: mg] — Population: one patient was missing
  mg
    number analyzed (Participants) | 67 | 63 | 130
    (all) | 20 [5 to 30.3] | 20 [7.5 to 25.3] | 20 [5 to 27]

OUTCOME MEASURES:

1. Primary Outcome: Residual Urine Volume
Description: Residual urine volume in the bladder as assessed by bladder scan
Time Frame: from Postoperative days 1 to POD 2 or until day of discharge whichever occurs first
Population: 17 patients were completely missing on urine residual. Multiple imputation was used solely for estimating the treatment effect on urinal residual. The summary statistics of urine residual for each day was reported based on original data.
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Treatment-Naloxegol | Placebo Arm
Number analyzed (Participants) | 59 | 55
ml
  Day 1 AM: number analyzed (Participants) | 40 | 46
  Day 1 AM | 62 [5 to 187] | 114 [13 to 247]
  Day 1 PM: number analyzed (Participants) | 41 | 43
  Day 1 PM | 48 [0 to 206] | 31 [0 to 169]
  Day 2 AM: number analyzed (Participants) | 39 | 39
  Day 2 AM | 32 [0 to 152] | 28 [0 to 122]
  Day 2 PM: number analyzed (Participants) | 32 | 37
  Day 2 PM | 0 [0 to 122] | 28 [0 to 66]
Statistical Analysis 1: Comparison: Treatment-Naloxegol; Test type: Superiority — multiple imputation for longitudinal data was conducted to impute the missing data for the primary outcome. The final results were obtained from pooling results from 10 imputed complete case data set; p = 0.84, Mixed Models Analysis; geometric mean ratio = 0.90, 95% CI 2-sided [0.32 to 2.55]
Statistical Analysis 2: Comparison: Treatment-Naloxegol vs Placebo Arm; Test type: Superiority — A sensitivity analysis using complete case analysis; p = 0.73, Mixed Models Analysis; geometric mean ratio = 0.82, 95% CI 2-sided [0.26 to 2.56]

2. Secondary Outcome: Side Effects of Naloxegol on Other Opioid Related Side Effects
Description: Opioid-related Symptom Distress Scale (ORSDS) is a 4 point-scale that evaluates three symptom distress dimensions (frequency, severity, bothersomeness) for opioid-related side effects. The 12 elements of the ORSDS are nausea, vomiting, constipation, difficulty passing urine, difficulty concentrating, drowsiness, lightheaded, fatigue, feeling confused, itchiness, dry mouth, and headache. The ORSDS questionnaire was administered by a trained investigator on first and second postoperative days while patients remained hospitalized. We reported the average ORSDS score from all 12 elements, which ranged from 0 to 4 and higher scores represent worse outcome.
Time Frame: Postoperative days 1-2 or until day of discharge whichever occurs first
Population: some patients were missing on this outcome at repeated measurements. A mixed effects model assuming auto-regressive correlation structure and the outcome was log-transformed
Measure: Median (Inter-Quartile Range); unit: log(score on a scale)
Arm/Group | Treatment-Naloxegol | Placebo Arm
Number analyzed (Participants) | 66 | 61
log(score on a scale)
  Day 1 | 0.53 [0.34 to 0.79] | 0.45 [0.31 to 0.81]
  Day 2: number analyzed (Participants) | 54 | 52
  Day 2 | 0.34 [0.2 to 0.64] | 0.34 [0.13 to 0.62]
Statistical Analysis 1: Comparison: Treatment-Naloxegol vs Placebo Arm; Test type: Superiority; p = 0.91, Mixed Models Analysis; geometric mean ratio = 1.02, 98.3% CI 2-sided [0.63 to 1.67]

3. Secondary Outcome: Need for Indwelling Urinary Catheterization
Description: Number of patients receiving Naloxegol requiring indwelling urinary catheters
Time Frame: Postoperative days 1-2 or until day of discharge whichever occurs first
Population: Our final analyzed study population had 131 patients since 5 patients did not complete (due to withdrawal or not receiving any treatment) the study thus were removed from the final analysis. Among 131 patients, 4 patients were missing from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment-Naloxegol | Placebo Arm
Number analyzed (Participants) | 65 | 62
Participants | 19 | 7
Statistical Analysis 1: Comparison: Treatment-Naloxegol vs Placebo Arm; Test type: Superiority; p = 0.012, Chi-squared; Risk Ratio (RR) = 2.58, 98.3% CI 2-sided [0.98 to 6.80]

4. Secondary Outcome: Quality of Recovery
Description: Quality of recovery is a validated scoring system that quantifies patients' early postoperative health status with range of 0-150 where higher score means better quality of recovery. We used the 15-question version, the QoR-15
Time Frame: Postoperative Days 2 or discharge day whichever was earlier
Population: We only had a total of 131 patients in our final analysis since 5 patients were removed from the final analysis due to not completing the study (withdrawal or not receiving any treatment). Among 131 patients, 9 patients were missing from this analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Treatment-Naloxegol | Placebo Arm
Number analyzed (Participants) | 63 | 59
units on a scale | 119 [103 to 131] | 123 [115 to 133]
Statistical Analysis 1: Comparison: Treatment-Naloxegol vs Placebo Arm; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney); median of differences = -5, 98.3% CI 2-sided [-12 to 2]

ADVERSE EVENTS:
Time Frame: until discharge from hospital, an average of 2 day, up to 3 days
Description: Adverse events of particular interest are:
  * Opioid withdrawal: hyperhidrosis, chills, diarrhea, abdominal pain, anxiety, irritability
  * Severe abdominal pain (>8/10) and/or diarrhea
  * Gastrointestinal perforation
Arm/Group | Treatment-Naloxegol | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/64
Serious Adverse Events (participants affected / at risk) | 1/67 | 0/64
Other Adverse Events (participants affected / at risk) | 0/67 | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment-Naloxegol (N=67) | Placebo Arm (N=64)
Troponin elevation and ST elevation (Cardiac disorders) | 1 (1) | 0 (0) — Patient was transferred to coronary ICU for further care. A heparin infusion was initiated. A left heart cath is planned for 5/31/2018. Reported to PI. Not related to study medication. Continue to follow patient status.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT03235739/Prot_SAP_006.pdf
  • Informed Consent Form (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT03235739/ICF_001.pdf